CLINICAL TRIAL: NCT04745988
Title: An Open Label Phase 2 Study to Evaluate the Safety and Efficacy of Lenvatinib with Pembrolizumab or Lenvatinib, Pembrolizumab and FLOT in the Neoadjuvant / Adjuvant Treatment for Patients with Gastric Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Center Hospital East (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Kohei Shitara, Chief of Gastroenterology and Gastrointestinal Oncology Division, National Cancer Center Hospital East
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPOC2001
Record Dates: First submitted 2021-02-08; First posted 2021-02-09 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — lenvatinib; pembrolizumab; Docetaxel; Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lenvatinib Plus Pembrolizumab (Experimental): One cycle is 21 days, with Lenvatinib plus Pembrolizumab repeated 3 cycles before surgery and 3 cycles after surgery, followed by 11 cycles of pembrolizumab monotherapy as the adjuvant treatment.
  Interventions: Drug: Lenvatinib 20mg; Drug: Pembrolizumab
- Lenvatinib, Pembrolizumab Plus FLOT (Experimental): One cycle is 21 days, with Lenvatinib, Pembrolizumab plus FLOT repeated 3 cycles before surgery and 3 cycles after surgery, followed by 11 cycles of pembrolizumab monotherapy as the adjuvant treatment.
  Interventions: Drug: Pembrolizumab; Drug: Lenvatinib 8mg; Drug: Docetaxel; Drug: Oxaliplatin; Drug: Levofolinate; Drug: Fluorouracil

INTERVENTIONS:
Drug: Lenvatinib 20mg — Lenvatinib will be administered at a dose of 20mg as oral dose, once a day.
  Arms: Lenvatinib Plus Pembrolizumab
Drug: Pembrolizumab — Pembrolizumab will be administered at a dose of 200mg as a 30-minutes IV infusion, Q3W (25 minutes to 40 minutes are acceptable).
Drug: Lenvatinib 8mg — Lenvatinib will be administered at a dose of 8mg as oral dose, once a day.
  Arms: Lenvatinib, Pembrolizumab Plus FLOT
Drug: Docetaxel — Docetaxel will be administered at a dose of 50mg/m^2 as a IV infusion, Q2W.
  Arms: Lenvatinib, Pembrolizumab Plus FLOT
Drug: Oxaliplatin — Oxaliplatin will be administered at a dose of 85mg/m^2 as a IV infusion, Q2W.
  Arms: Lenvatinib, Pembrolizumab Plus FLOT
Drug: Levofolinate — Levofolinate will be administered at a dose of 200mg/m^2 as a IV infusion, Q2W.
  Arms: Lenvatinib, Pembrolizumab Plus FLOT
Drug: Fluorouracil — Levofolinate will be administered at a dose of 2600mg/m^2 as a IV infusion, Q2W.
  Arms: Lenvatinib, Pembrolizumab Plus FLOT

SUMMARY:
This study is an open label phase 2 study to evaluate the safety and efficacy of Lenvatinib with Pembrolizumab or Lenvatinib, Pembrolizumab and FLOT in the neoadjuvant / adjuvant treatment for Patients with Gastric Cancer.

DETAILED DESCRIPTION:
This study is an open-label, single-arm, single-center, phase 2 clinical trial. Eligible patients are with previously untreated gastric and gastroesophageal junction adenocarcinoma as defined by cT2-4 and/or cN+ without evidence of metastatic disease. Patients in the exploratory cohort will receive 3 cycles of 20 mg oral Lenvatinib daily plus 200 mg intravenous Pembrolizumab every 3 weeks as the neoadjuvant treatment followed by surgery, and then 3 cycles of Lenvatinib plus Pembrolizumab followed by 11 cycles of Pembrolizumab monotherapy as the adjuvant treatment. Also, Patients in the FLOT cohort will receive 3 cycles of 8 mg oral Lenvatinib daily, 200 mg intravenous Pembrolizumab every 3 weeks and FLOT (Docetaxel 50 mg/m2, Oxaloplatin 85 mg/m2, Levofolinate 200 mg/m2, 5-FU 2600 mg/m2) every 2 weeks as the neoadjuvant treatment followed by surgery, and then 3 cycles of Lenvatinib ,Pembrolizumab plus FLOT followed by 11 cycles of Pembrolizumab monotherapy as the adjuvant treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Have gastric and gastroesophageal junction adenocarcinoma
2. Untreated and cT2-4 and/or cN+ without evidence of metastatic disease
3. Patients at least 20 years of age on the day of providing consent.
4. Patients with a performance status of 0 or 1 on the Eastern Cooperative Oncology Group.
5. Patients with adequate organ function at the time of enrollment as defined below:

   * Neutrophil count ≥1500mm3
   * Platelet count ≥10 × 100,000/mm3
   * Hemoglobin (Hb) ≥ 9.0 g/dL,
   * Total bilirubin ≤1.5 mg/dL
   * AST (GOT) and ALT (GPT) ≤ 100 IU/L
   * Creatinine ≤1.5 mg/dL
   * Urinary protein : It satisfies one of the following (if any of the inspection criteria are satisfied, other examination may not be carried out) (i) urinary protein (test paper method) is 2+ or less (ii) Urine Protein Creatinine (UPC) ratio <3.5 (iii) 24-hour urine protein was measured, urinary protein ≦ 3500 mg
   * International normalized ratio (INR) ≤ 1.5
6. Patients who not received a blood transfusion within 14 days of registration.
7. Patients have recovered adverse events associated with radiation and surgical operation as pretreatment to Grade 1 or less or baseline or less with CTCAE v5.0 excluding stable symptoms. However, adverse events with stable symptoms even with Grade 2 or higher excluded.
8. Female of childbearing potential who are negative in a pregnancy test within 14 days before enrollment. Both male and female patients should agree to use an adequate method of contraception (total abstinence or use of a male condom plus partner use of contraceptive method [an intrauterine device or hormone releasing system, a contraceptive implant and an oral contraceptive]) starting with the first dose of study therapy through 120 days after the last dose of study therapy. Duration will be determined when the subject is assigned to treatment.
9. Patients capable of taking oral medication.
10. Patients who provided written informed consent to be subjects in this study.

Exclusion Criteria:

1. Patients who have undergone surgical treatment and radiotherapy within 2 weeks before enrollment.
2. Patients with hypertension that is difficult to control (systolic blood pressure ≥160 mmHg and diastolic blood pressure ≥90 mmHg) despite treatment with several hypotensive agents.
3. Patients with acute coronary syndrome (including myocardial infarction and unstable angina), and with a history of coronary angioplasty or stent placement performed within 6 months before enrollment.
4. Patients with a history of New York Heart Association congestive heart failure of grade II or above, unstable angina, myocardial infarction.
5. Patients have an addigional active malignancy (except for definitively treated melanoma in-situ, basal or squamous cell carcinoma of the skin, or carcinoma in-situ of the cervix) within the past 24 months.
6. Patients have severe (hospitalization required) complications (intenstinal palsy, intestinal obstruction, pulmonary fibrosis, diabetes difficult to control, heart failure, myocardial infarction, unstable angina, renal failure, liver failure, mental disease, cerebrovascular disease etc).
7. Patients with a history of a gastrointestinal perforation and /or gastrointestinal fistula within 6 months before enrollment.
8. Is infected with active hepatitis B (defined as HBs antigen positive) or hepatitis C.
9. Patients with a history of human immunodeficiency virus (HIV).
10. Patients with a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
11. Patients who are administered live vaccines <30 days before the initiation of treatment with the investigational drug.
12. Patients with concurrent autoimmune disease, or a history of chronic or recurrent autoimmune disease.
13. Patients who require systemic corticosteroids (excluding temporary usage for tests, prophylactic administration for allergic reactions, or to alleviate swelling associated with radiotherapy) or immunosuppressants, or who have received such a therapy <14 days before enrollment.
14. Patients have serious non-healing wound, ulcer, or bone fracture.
15. Females who are pregnant or breastfeeding.
16. Patients have no intention to comply with the protocol or cannot comply.
17. Patients were judged unsuitable as subject of this study by investigator.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2021-11-11 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Major pathological response (MPR) rate | 6 months
  The MPR rate will be defined as the proportion of patients whose percentage of residual tumor in the stomach and lymph node decreased to < 10%, as determined by a pathologist.

SECONDARY OUTCOMES:
Pathological complete response (pCR) rate | 6 months
  The pCR rate will be defined as the proportion of patients whose tumor in the stomach and lymph node completely disappeared, as determined by a pathologist.
Tumor response in the gastric primary lesion | 6 months
  The number of patients achieving endoscopic CR, PR, SD, or PD will be separately tabulated.
Radical resection rate | 6 months
  The radical resection rate will be defined as the proportion of patients who underwent a radical resection (R0 resection).
Treatment completion rate until surgery | 6 months
  The treatment completion rate will be defined as the proportion of patients who started the protocol treatment, completed a three-cycle treatment with the study drug, and then underwent a radical resection (R0 resection).
Treatment completion rate until adjuvant treatment | 1 year 8 months
  The treatment completion rate will be defined as the proportion of patients who started the protocol treatment, completed a three-cycle treatment with the study drug, and then underwent a radical resection (R0 resection) and adjuvant treatment was performed up to 14 cycles.
Event free survival (EFS) | 3 years
  The registration date is the starting date, and is defined as the period until the event that occurs any of the following.
  * Disease progression based on image evaluation using RECIST 1.1
  * Recurrence based on CT or biopsy among patients with no postoperative lesions
  * Death of any cause If it is determined to be exacerbated based on the image evaluation, the inspection date on which the image inspection was performed shall be the exacerbation date.
  Secondary primary malignancies are not an EFS event. Patients for whom no EFS event has been recorded will be censored on the final image evaluation date.
Overall survival (OS) | 3 years
  The period will be from the day of enrollment, as the starting date of the computation, to the day of death of any cause.
  Surviving patients should be censored on the last day of PFS confirmed (Confirmation of survival by telephone inquiry will be acceptable. However, the fact of confirming survival should be documented in medical records.).
  Patients who are lost to follow up should be censored on the last day when their survival is confirmed before being lost to follow up.
The incidence of adverse events | Up to 30 days after the last dose
  For adverse events due to protocol treatment, determine the frequency of worst grades in all courses according to CTCAE v5.0, the incidence of adverse events of Grade 3 or higher, and the incidence of adverse events of Grade 4 or higher.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center Hospital East, Kashiwa, Chiba, Japan

IPD SHARING:
Plan to Share IPD: No